CLINICAL TRIAL: NCT01956110
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre, Multinational Trial Comparing the Efficacy and Safety of FE 999049 With Follitropin Alfa (GONAL-F) in Controlled Ovarian Stimulation in Women Undergoing an Assisted Reproductive Technology Programme
Brief Title: Evidence-based Stimulation Trial With Human rFSH in Europe and Rest of World 1
Acronym: ESTHER-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000004; 2013-001669-17 (EudraCT Number); U1111-1147-6826 (Other: WHO)
Record Dates: First submitted 2013-08-16; First posted 2013-10-08 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2018-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta; FE 999049; follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Follitropin Delta (FE 999049)
  Interventions: Drug: Follitropin Delta (FE 999049)
- B (Active Comparator): Follitropin Alfa (GONAL-F)
  Interventions: Drug: Follitropin Alfa (GONAL-F)

INTERVENTIONS:
Drug: Follitropin Delta (FE 999049)
  Arms: A
Drug: Follitropin Alfa (GONAL-F)
  Arms: B

SUMMARY:
This trial investigates the effects of FE 999049 compared to GONAL-F.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Documents signed prior to screening evaluations
* In good physical and mental health
* Pre-menopausal females between the ages of 18 and 40 years
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II or with partners diagnosed with male factor infertility, eligible for in vitro fertilisation (IVF) and/or intracytoplasmic sperm injection (ICSI) using fresh or frozen ejaculated sperm from male partner or sperm donor
* Infertility for at least one year before randomisation for subjects ≤37 years or for at least 6 months for subjects ≥38 years (not applicable in case of tubal or severe male factor infertility)
* The trial cycle will be the subject's first controlled ovarian stimulation cycle for IVF/ICSI
* Hysterosalpingography, hysteroscopy, saline infusion sonography, or transvaginal ultrasound documenting a uterus consistent with expected normal function (e.g. no evidence of clinically interfering uterine fibroids defined as submucous or intramural fibroids larger than 3 cm in diameter, no polyps and no congenital structural abnormalities which are associated with a reduced chance of pregnancy) within 1 year prior to randomisation
* Transvaginal ultrasound documenting presence and adequate visualisation of both ovaries, without evidence of significant abnormality (e.g. no endometrioma greater than 3 cm or enlarged ovaries which would contraindicate the use of gonadotropins) and normal adnexa (e.g. no hydrosalpinx) within 1 year prior to randomisation. Both ovaries must be accessible for oocyte retrieval.
* Early follicular phase (cycle day 2-4) serum levels of FSH between 1 and 15 IU/L (results obtained within 3 months prior to randomisation)
* Body mass index (BMI) between 17.5 and 32.0 kg/m2 (both inclusive) at screening

Exclusion Criteria:

* Known endometriosis stage III-IV
* One or more follicles ≥10 mm observed on the transvaginal ultrasound prior to randomisation on stimulation day 1
* Known history of recurrent miscarriage (defined as three consecutive losses after ultrasound confirmation of pregnancy (excl. ectopic pregnancy) and before week 24 of pregnancy)
* Known abnormal karyotype of subject or of her partner/sperm donor, as applicable, depending on source of sperm used for insemination in this trial.
* Any known clinically significant systemic disease (e.g. insulin-dependent diabetes)
* Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) which can compromise participation in the trial with the exception of controlled thyroid function disease
* Known tumours of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus which would contraindicate the use of gonadotropins.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1329 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (13):
- UZ Brussel (there may be other sites in this country), Brussels, Belgium
- Fertilitat and PUC-RS (there may be other sites in this country), Porto Alegre, Brazil
- Canada (3):
  - Pacific Centre for Reproductive Medicine, Burnaby, British Columbia
  - Olive Fertility Centre, Vancouver, British Columbia
  - Ottawa Fertility Centre, Ottawa, Ontario
- IVF CUBE SE (there may be other sites in this country), Prague, Czechia
- Rigshospitalet Fertilitetsklinikken (there may be other sites in this country), Copenhagen, Denmark
- Department of Endocrine Gynaecology and Reproductive Medicine, Hôpital Jeanne de Flandre (there may be other sites in this country), Lille, France
- Centro Natalità San Raffaele (there may be other sites in this country), Milan, Italy
- The nOvum Clinic (there may be other sites in this country), Warsaw, Poland
- IVF & Reproductive Genetics Center (there may be other sites in this country), Moscow, Russia
- IVI Sevilla (there may be other sites in this country), Seville, Spain
- Glasgow Centre for Reproductive Medicine Ltd. (there may be other sites in this country), Glasgow, United Kingdom

REFERENCES:
- [Result] Arce JC, Larsson P, Garcia-Velasco JA. Establishing the follitropin delta dose that provides a comparable ovarian response to 150 IU/day follitropin alfa. Reprod Biomed Online. 2020 Oct;41(4):616-622. doi: 10.1016/j.rbmo.2020.07.006. Epub 2020 Jul 15. PMID 32819842
- [Result] Havelock J, Aaris Henningsen AK, Mannaerts B, Arce JC; ESTHER-1 and ESTHER-2 Trial Groups. Pregnancy and neonatal outcomes in fresh and frozen cycles using blastocysts derived from ovarian stimulation with follitropin delta. J Assist Reprod Genet. 2021 Oct;38(10):2651-2661. doi: 10.1007/s10815-021-02271-5. Epub 2021 Jul 13. PMID 34254211
- [Result] Ishihara O, Nelson SM, Arce JC. Comparison of ovarian response to follitropin delta in Japanese and White IVF/ICSI patients. Reprod Biomed Online. 2022 Jan;44(1):177-184. doi: 10.1016/j.rbmo.2021.09.014. Epub 2021 Sep 23. PMID 34799275
- [Derived] Nelson SM, Larsson P, Mannaerts BMJL, Nyboe Andersen A, Fauser BCJM. Anti-Mullerian hormone variability and its implications for the number of oocytes retrieved following individualized dosing with follitropin delta. Clin Endocrinol (Oxf). 2019 May;90(5):719-726. doi: 10.1111/cen.13956. Epub 2019 Mar 18. PMID 30801744
- [Derived] Nyboe Andersen A, Nelson SM, Fauser BC, Garcia-Velasco JA, Klein BM, Arce JC; ESTHER-1 study group. Individualized versus conventional ovarian stimulation for in vitro fertilization: a multicenter, randomized, controlled, assessor-blinded, phase 3 noninferiority trial. Fertil Steril. 2017 Feb;107(2):387-396.e4. doi: 10.1016/j.fertnstert.2016.10.033. Epub 2016 Nov 29. PMID 27912901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 sites randomised subjects into the trial : 3 in Belgium, 3 in Brazil, 3 in Canada, 4 in the Czech Republic, 2 in Denmark, 2 in France, 2 in Italy, 2 in Poland, 4 in Russia, 10 in Spain and 2 in United Kingdom.
Pre-assignment Details: A total of 1501 subjects were screened in the trial, of whom 1329 subjects were randomised: 666 subjects to FE 999049 and 663 subjects to GONAL-F. Three subjects were randomisation failures and did not receive investigational medicinal product (IMP); 1 in the FE 999049 group and 2 in the GONAL-F group.
Groups:
- FE 999049: FE 999049 was administered as single daily subcutaneous injections in the abdomen. Subjects randomised to FE 999049 had their individual dose determined on the basis of their anti-Müllerian hormone (AMH) level at screening and their body weight at randomisation. The daily FE 999049 dose was fixed throughout the stimulation period and maximum allowed daily dose was 12 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Subjects could be treated for a maximum of 20 days.
- GONAL-F: Follitropin Alfa (GONAL-F) was administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F was 150 international units (IU) and fixed for the first five stimulation days, after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Subjects could be treated for a maximum of 20 days.
Period: Overall Study
Arm/Group | FE 999049 | GONAL-F
Started | 665 | 661
Completed | 630 | 639
Not Completed | 35 | 22
Not completed — Protocol Violation | 25 | 11
Not completed — Adverse Event | 9 | 10
Not completed — Personal reasons | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of the 1,329 randomised subjects, 1,326 were exposed to IMP: FE 999049 (665 subjects) and GONAL-F (661 subjects). The 3 subjects who were not exposed to IMP were randomisation failures; 2 subjects (1 in each treatment group) did not fulfil an inclusion criterion, and 1 subject (in the GONAL-F group) withdrew due to personal reasons.
Groups:
- FE 999049: FE 999049 was administered as single daily subcutaneous injections in the abdomen. Subjects randomised to FE 999049 had their individual dose determined on the basis of their AMH level at screening and their body weight at randomisation. The daily FE 999049 dose was fixed throughout the stimulation period and maximum allowed daily dose was 12 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Subjects could be treated for a maximum of 20 days.
- GONAL-F: GONAL-F was administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F was 150 IU and fixed for the first five stimulation days, after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Subjects could be treated for a maximum of 20 days.
- Total: Total of all reporting groups
Arm/Group | FE 999049 | GONAL-F | Total
Number analyzed (Participants) | 665 | 661 | 1326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 665 | 661 | 1326
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 665 | 661 | 1326
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate
Description: Ongoing pregnancy was defined as at least one intrauterine viable fetus 10-11 weeks after blastocyst transfer.
Time Frame: 10-11 weeks after blastocyst transfer
Population: Modified intention-to-treat (mITT) analysis set (all randomised and exposed subjects). This is equivalent to full analysis set (FAS).
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects | 30.7 | 31.6
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; The pre-specified non-inferiority margin was -8.0% (absolute). Non-inferiority was evaluated based on a two-sided 95% confidence interval (CI) derived based on the asymptotic normal distribution. The treatment comparison was adjusted for age (<35, 35-37 and 38-40 years) by using the Mantel-Haenszel method to combine results across age-strata; Test type: Non-Inferiority — The lower bound of the 95% CI was well above the pre-specified non-inferiority limit of -8.0%. Thus, non-inferiority of FE 999049 to GONAL-F with regard to ongoing pregnancy rate was demonstrated; Treatment difference = -0.9, 95% CI 2-sided [-5.9 to 4.1]

2. Primary Outcome: Ongoing Implantation Rate
Description: Ongoing implantation rate was defined as the number of intrauterine viable fetuses 10-11 weeks after transfer divided by number of blastocysts transferred.
Time Frame: 10-11 weeks after blastocyst transfer
Population: Subjects with blastocyst transfer (a total of 585 and 584 blastocysts were transferred in the FE999049 and GONAL-F groups, respectively).
Measure: Number; unit: Percentage
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 562 | 560
Percentage | 35.2 | 35.8
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; The pre-specified non-inferiority margin was -8.0% (absolute). Non-inferiority was evaluated based on a two-sided 95% CI derived based on the asymptotic normal distribution. The treatment comparison was adjusted for age (<35, 35-37 and 38-40 years) by using the Mantel-Haenszel method to combine results across age-strata; Test type: Non-Inferiority — The lower bound of the 95% CI was well above the pre-specified non-inferiority limit of -8.0%. Thus, non-inferiority of FE 999049 to GONAL-F with regard to ongoing implantation rate was demonstrated; Treatment difference = -0.6, 95% CI 2-sided [-6.1 to 4.8]

3. Secondary Outcome: Vital Pregnancy Rate
Description: Vital pregnancy was defined as at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after blastocyst transfer.
Time Frame: 5-6 weeks after blastocyst transfer
Population: mITT analysis set (all randomised and exposed subjects). This is equivalent to the FAS.
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects | 31.7 | 33.4
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment groups were compared using a two-sided 95% CI derived based on the asymptotic normal distribution. The treatment comparison was adjusted for age (<35, 35-37 and 38-40 years) by using the Mantel-Haenszel method to combine results across age-strata; Test type: Non-Inferiority — The lower bound of the 95% CI was well above -8.0% (pre-specified non-inferiority limit for the co-primary endpoints). Thus, the result was supportive of the co-primary endpoint analyses; Treatment difference = -1.6, 95% CI 2-sided [-6.7 to 3.4]

4. Secondary Outcome: Implantation Rate
Description: Implantation rate was defined as the number of gestational sacs 5-6 weeks after transfer divided by number of blastocysts transferred.
Time Frame: 5-6 weeks after blastocyst transfer
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 562 | 560
Percentage | 39.8 | 41.3
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Treatment difference = -1.4, 95% CI 2-sided [-7.0 to 4.2]

5. Secondary Outcome: Proportion of Subjects With Extreme Ovarian Responses, Defined as <4, ≥15 or ≥20 Oocytes Retrieved
Time Frame: Day of oocyte retrieval
Population: Subjects who underwent triggering of final follicular maturation.
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 635 | 643
Percentage of subjects
  <4 or >=15 oocytes retrieved | 26.6 | 31.3
  <4 or >=20 oocytes retrieved | 14.5 | 18.4
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: <4 or >=15 oocytes retrieved; Test type: Other — A logistic regression model was fitted to the data including AMH, log(AMH)^2, treatment group and interactions between treatment group and AMH and treatment group and log(AMH)^2 in the linear predictor. A second logistic regression model (nested within the first model) was fitted including AMH and log(AMH)^2 in the linear predictor; p = 0.001, Likelihood ratio test — Inclusion of treatment provides a better fit to the data; Likelihood ratio test comparing the reduced model including only AMH to the full model including AMH, treatment group and interactions
Statistical Analysis 2: Comparison: FE 999049 vs GONAL-F; Treatment comparison: <4 or >=20 oocytes retrieved; Test type: Other — A logistic regression model was fitted to the data including AMH, log(AMH)2, treatment group and interactions between treatment group and AMH and treatment group and log(AMH)^2 in the linear predictor. A second logistic regression model (nested within the first model) was fitted including AMH and log(AMH)^2 in the linear predictor; p = 0.002, Likelihood ratio test — Inclusion of treatment provides a better fit to the data; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Proportion of Subjects With Early OHSS (Ovarian Hyperstimulation Syndrome) and/or Preventive Interventions for Early OHSS
Description: The proportion of subjects with early OHSS, early OHSS of moderate or severe grade, preventive interventions for early OHSS, early OHSS and/or preventive interventions for early OHSS, and early OHSS of moderate or severe grade and/or preventive interventions for early OHSS are presented.
Time Frame: ≤9 days after triggering of final follicular maturation
Population: mITT analysis set (all randomised and exposed subjects). This is equivalent to the FAS.
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects
  Early OHSS (any grade) | 2.6 | 3.0
  Early OHSS (moderate/severe) | 1.4 | 1.4
  Any preventive intervention | 2.3 | 4.5
  Early OHSS (any grade) / preventive interventions | 4.7 | 6.2
  Early OHSS (mod/severe) / preventive interventions | 3.6 | 5.1
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Early OHSS (any grade); Test type: Other — Nested logistic regression models were compared using the likelihood ratio test. The full logistic regression model included treatment as factor, log(AMH) as covariate and the interaction term. The nested model did not include treatment and the interaction term; p = 0.291, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Early OHSS (moderate/severe); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.644, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Preventive interventions; Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.005, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Early OHSS (any grade) and/or preventive interventions; Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.046, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Early OHSS (moderate/severe) and/or preventive interventions; Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.019, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]

7. Secondary Outcome: Proportion of Subjects With Cycle Cancellation Due to Poor Ovarian Response or Excessive Ovarian Response
Description: Proportion of subjects with cycle cancellation due to poor ovarian response, excessive ovarian response, and triggering with gonadotropin-releasing hormone (GnRH) agonist are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: mITT analysis set (all randomised and exposed subjects). This is equivalent to the FAS.
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects
  Cycle cancelled due to poor ovarian response | 3.8 | 2.7
  Cycle cancelled due to excessive ovarian response | 0 | 0
  Triggering with GnRH agonist | 1.5 | 3.5
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Cycle cancelled due to poor response; Test type: Equivalence — Treatment groups were compared using a logistic regression model with treatment and age (<35, 35- 37, and 38-40 years) as factors; p = 0.302, Likelihood ratio test — P-value corresponds to test for treatment difference; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.74 to 2.57]
Statistical Analysis 2: Comparison: FE 999049 vs GONAL-F; Treatment comparison:Triggering with GnRH agonist; Test type: Equivalence — Treatment groups were compared using a logistic regression model with treatment and age (<35, 35-37, and 38-40 years) as factors; p = 0.019, Likelihood ratio test — P-value corresponds to test for treatment difference; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.2 to 0.9]

8. Secondary Outcome: Number of Oocytes Retrieved
Time Frame: Day of oocyte retrieval
Population: Subjects who underwent triggering of final follicular maturation.
Measure: Mean (Standard Deviation); unit: Oocytes retrieved
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 636 | 643
Oocytes retrieved | 10.0 (5.6) | 10.4 (6.5)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Number of oocytes retrieved; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.692, van Elteren

9. Secondary Outcome: Proportion of Subjects With <4, 4-7, 8-14, 15-19 and ≥20 Oocytes Retrieved
Time Frame: Day of oocyte retrieval
Population: Subjects who underwent triggering of final follicular maturation.
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 635 | 643
Percentage of subjects
  Low response (<4 oocytes) | 8.0 | 9.6
  Moderate response (4-7 oocytes) | 30.1 | 30.3
  Targeted response (8-14 oocytes) | 43.3 | 38.4
  Hyperresponse (15-19 oocytes) | 12.1 | 12.9
  Severe hyperresponse (≥ 20 oocytes) | 6.5 | 8.7
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; The relation between ovarian response potential (AMH at screening) and probability of achieving the targeted response was modelled using logistic regression models; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.019, Likelihood ratio test — Inclusion of treatment provides a better fit to the data; [statistical method as in outcome 5, analysis 1]

10. Secondary Outcome: Percentage of Metaphase II Oocytes (Oocytes Inseminated Using ICSI [Intracytoplasmic Sperm Injection])
Description: Number of oocytes in metaphase II prior to ICSI insemination is presented.
Time Frame: Prior to insemination
Population: Subjects with all oocytes inseminated using ICSI.
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 531 | 522
Number of oocytes | 7.4 (4.3) | 7.7 (5.2)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Number of metaphase II oocytes; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.909, van Elteren

11. Secondary Outcome: Fertilisation Rate
Description: Fertilisation rate was defined as the number of oocytes with 2 pronuclei divided by the number of oocytes retrieved.
Time Frame: Day 1 after insemination
Population: Subjects with oocytes retrieved.
Measure: Mean (Standard Deviation); unit: Percentage of oocytes
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 634 | 640
Percentage of oocytes | 56 (24.5) | 57 (23.8)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Fertilisation rate; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.53, van Elteren

12. Secondary Outcome: Number and Quality of Embryos on Day 3
Description: Number of embryos (total and good-quality) on Day 3 are presented. A good-quality embryo was defined as an embryo with ≥6 blastomeres and fragmentation ≤20% on Day 3.
Time Frame: On day 3 after oocyte retrieval
Population: Subjects with oocytes retrieved.
Measure: Mean (Standard Deviation); unit: Number of embryos
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 634 | 640
Number of embryos
  Number of embryos | 5.4 (3.7) | 5.7 (4.3)
  Number of good-quality embryos | 4.2 (3.3) | 4.5 (3.7)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Number of embryos; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.59, van Elteren
Statistical Analysis 2: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Good quality embryos; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.414, van Elteren

13. Secondary Outcome: Number and Quality of Blastocysts on Day 5
Description: Number of blastocysts (total and good-quality) on Day 5 are presented. A good-quality blastocyst was defined as a blastocyst of grade 3BB or higher.
Time Frame: On day 5 after oocyte retrieval
Population: Subjects with oocytes retrieved.
Measure: Mean (Standard Deviation); unit: Number of blastocytss
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 634 | 640
Number of blastocytss
  Number of blastocysts | 3.3 (2.8) | 3.5 (3.2)
  Number of good-quality blastocysts | 2.0 (2.2) | 2.1 (2.4)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Number of blastocysts; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.344, van Elteren
Statistical Analysis 2: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Good-quality blastocysts; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.58, van Elteren

14. Secondary Outcome: Total Gonadotropin Dose
Description: The total gonadotropin dose was recorded.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: mITT analysis set (all randomised and exposed subjects). This is equivalent to the FAS.
Measure: Mean (Standard Deviation); unit: µg of dose
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
µg of dose | 90 (25.3) | 103.7 (33.6)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Total gonadotropin dose; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p < 0.001, van Elteren

15. Secondary Outcome: Number of Stimulation Days
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: mITT analysis set (all randomised and exposed subjects). This is equivalent to the FAS.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Days | 8.9 (1.9) | 8.6 (1.7)
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Number of stimulation days; Test type: Equivalence — Treatment groups were compared using the van Elteren test adjusted for age (<35, 35-37, and 38-40 years); p = 0.062, van Elteren

16. Secondary Outcome: Proportion of Subjects With Investigator-requested Gonadotropin Dose Adjustments
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: mITT analysis set (all randomised and exposed subjects). This is equivalent to the FAS.
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects | 33.2 | 36.8
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Investigator-requested gonadotropin dose adjustments; Test type: Equivalence — Treatment groups were compared using a chi-square test; p = 0.178, Chi-squared

17. Secondary Outcome: Frequency of Injection Site Reactions (Redness, Pain, Itching, Swelling and Bruising) Assessed by the Subject During the Stimulation Period
Description: Subjects self-assessed injection site reactions (redness, itching, pain, swelling and bruising) immediately, 30 minutes and 24 hours after each injection. The injection site reactions were assessed as none, mild, moderate and severe. The frequency of injection site reactions (mild, moderate or severe) based on all assessments performed is presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Number; unit: Percentage of events
Groups:
- GONAL-F: GONAL-F was administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F was 150 IU and fixed for the first five stimulation days, after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Subjects could be treated for a maximum of 20 days.
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of events | 3.4 | 3.5

18. Secondary Outcome: Abdominal Discomfort Related to Controlled Ovarian Stimulation as Assessed by a Visual Analogue Scale (VAS)
Description: The subject self-assessed abdominal discomfort related to controlled ovarian stimulation using a VAS going from 0 mm (no abdominal discomfort) to 100 mm (worst imaginable abdominal discomfort).
Time Frame: End-of-stimulation and day of blastocyst transfer
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Millimeter
  End of stimulation visit | 16.1 (18.14) | 15.9 (17.36)
  Transfer visit | 17.2 (20.02) | 16.1 (19.37)

19. Secondary Outcome: Changes in Body Weight
Description: Change in body weight from baseline to end-of-stimulation and from baseline to day of blastocyst transfer.
Time Frame: End-of-stimulation and day of blastocyst transfer
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Kg
  End of stimulation visit | 0.3 (1.11) | 0.2 (0.78)
  Transfer visit | 0.0 (1.03) | 0.0 (0.98)

20. Secondary Outcome: Changes in Maximum Abdominal Circumference
Description: Change in maximum abdominal circumference from baseline to end-of-stimulation and from baseline to day of blastocyst transfer.
Time Frame: End-of-stimulation and day of blastocyst transfer
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Centimeter
  End of stimulation visit | 0.3 (4.41) | 0.1 (5.03)
  Transfer visit | 0.6 (4.79) | -0.1 (5.23)

21. Secondary Outcome: Proportion of Subjects With Treatment-induced Anti-follicle-stimulating Hormone (FSH) Antibodies
Description: The proportion of subjects with at least one treatment-induced anti-FSH antibody response at any time point.
Time Frame: Stimulation day 1, 7-10 days after last FE 999049 or GONAL-F dose and 21-28 days after last FE 999049 or GONAL-F dose
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects | 1.05 [0.42 to 2.16] | 0.76 [0.25 to 1.76]

22. Secondary Outcome: Proportion of Subjects With Late OHSS
Description: Late OHSS was defined as OHSS with onset >9 days after triggering of final follicular maturation.The proportion of subjects with late OHSS, and late OHSS of moderate or severe grade are presented.
Time Frame: >9 days after triggering of final follicular maturation
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects
  Late OHSS (any grade) | 0.9 | 1.8
  Late OHSS (moderate/severe) | 0.8 | 1.5
Statistical Analysis 1: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Late OHSS (any grade); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.320, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: FE 999049 vs GONAL-F; Treatment comparison: Late OHSS (moderate/severe); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.390, Likelihood ratio test — Inclusion of treatment does not provide a better fit to the data; [statistical method as in outcome 5, analysis 1]

23. Secondary Outcome: Technical Malfunctions of the Administration Pen
Description: Confirmed technical malfunction of administration pen.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: Safety analysis set (all randomised and exposed subjects). This is equivalent to the mITT (FAS).
Measure: Number; unit: Percentage of subjects
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 665 | 661
Percentage of subjects | 0.15 | 0.00

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from signed informed consent to the end-of-trial (up to approximately 5.5 months).
Description: AEs with onset after start of first administration of IMP were considered treatment-emergent and are presented for the safety analysis set.
Arm/Group | FE 999049 | GONAL-F
Serious Adverse Events (participants affected / at risk) | 16/665 | 10/661
Other Adverse Events (participants affected / at risk) | 168/665 | 159/661
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (N=665) | GONAL-F (N=661)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 3 (3) | 6 (6)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (N=665) | GONAL-F (N=661)
Procedural pain (Injury, poisoning and procedural complications) | 49 (51) | 52 (54)
Headache (Nervous system disorders) | 97 (131) | 88 (110)
Pelvic pain (Reproductive system and breast disorders) | 46 (54) | 41 (59)
Pelvic discomfort (Reproductive system and breast disorders) | 38 (46) | 25 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.